CLINICAL TRIAL: NCT03320694
Title: Comparison of Metformin and Insulin for Management of Gestational Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, Professor Obs Gynae, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/2015/211/SIMS
Record Dates: First submitted 2017-09-30; First posted 2017-10-25 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
Keywords: Gestational Diabetes Mellitus, Metformin, Insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Metformin; Insulin; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin (Experimental): Metformin will be given until 2500mg in divided doses till normoglycemia is achieved and will be continued till delivery
  Interventions: Drug: Metformin
- Insulin (Active Comparator): Insulin will be give as 3 regular injection and one intermediate acting injection at bedtime till normoglycemia is achieved and will be continued till delivery
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — metformin 500mg twice daily & increased until 2500mg till normoglycemia was achieved and was continued till delivery
  Other Names: Glucophage
  Arms: metformin
Drug: Insulin — The insulin group was given 3 S/C injections of regular insulin & one intermediate acting injection at night till normoglycemia was achieved and was continued till delivery
  Other Names: Humulin R U 100 and Humulin N
  Arms: Insulin

SUMMARY:
Gestational diabetic mellitus (GDM) patients randomised to metformin or insulin group.Aim was to achieve blood sugar levels of Blood sugar fasting (BSF) <5.3 mmol/l and 1 hour post meal<7.8mmol/l. Both groups were followed till delivery and outcome studied.

DETAILED DESCRIPTION:
75 gm Oral Glucose Tolerance Test (OGTT) was done in pregnant patients. Blood sugar fasting(BSF) > 5.5 mmol/l & 2 hours postprandial >7.8 mmol/l was labelled as GDM. They were randomised to metformin or insulin group. Those assigned to metformin group were started metformin 500mg twice daily & increased until 2500mg depending on the blood sugar levels. Aim was to achieve blood sugar levels of BSF <5.3 mmol/l and 1 hour post meal<7.8mmol/l. If blood sugar levels were not controlled, insulin was added. The insulin group was given 3 injections of regular insulin & one intermediate acting insulin injection at night subcutaneously. Both groups were followed till delivery and outcome studied

ELIGIBILITY:
Inclusion Criteria:•

* All pregnant Diagnosed GDM in pregnancy by OGTT from 22 week to 34 week with singleton pregnancy

Exclusion Criteria:

* Patients with Known diabetes mellitus
* Patients with multiple pregnancy
* With essential hypertension or pre eclampsia
* Patients having fetal malformation incompatible with life
* Patients with intrauterine death of fetus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
maternal glycemic control | From time of randomisation till 40 weeks
  Maternal glycemic control was measured by blood sugar levels

SECONDARY OUTCOMES:
Fetal macrosomia | at birth
  Birth weight more than 4kg
Apgar score | at birth
  <7 at 5min
Neonatal intensive care unit (NICU) stay | >24 hours after birth
  Admitted to NICU
Perinatal death | 7 days of delivery
  Fetal or neonatal death within 7 days
mode of delivery | at delivery
  Lower segment cesarean section , Spontaneous Vaginal Delivery, Instrumental delivery
Neonatal hypoglycemia | at birth
  Neonatal blood sugar was checked at birth and if <2.2mmol/l, was labelled

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan